CLINICAL TRIAL: NCT05307276
Title: Limitation of the Ventilatory Response to Exercise in the Master Athlete: Influences on Locomotor Muscle Fatigue and on Endurance Performance
Brief Title: Limitation of the Ventilatory Response to Exercise in the Master Athlete
Acronym: LAHMESS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Organisation problem
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 21-PP-10
Record Dates: First submitted 2022-03-08; First posted 2022-04-01 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — heliox; Air

STUDY DESIGN:
Intervention Model Description: Following the selection visit (#V0) to verify the inclusion and non-inclusion criteria, participants will make 2 visits (#V1 and #V2) including in particular a Respiratory Functional Exploration (EFR) and a triangular VO2 MAX estimation test in Ambient Air or Heliox conditions (depending on randomization).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy volunteers (Other): Following the selection visit (#V0) to verify the inclusion and non-inclusion criteria, participants will make 2 visits (#V1 and #V2) including in particular a Respiratory Functional Exploration (EFR) and a triangular
  Interventions: Other: Heliox; Other: Air

INTERVENTIONS:
Other: Heliox — Participants will then complete 1 FAM (#V3) to Neuromuscular Function Assessment (PRE-POST), Pre- and Post- Exercise Ventilatory Function Assessment, and a Constant Load Ergocycle Test to Tolerance Limit (intensity fixed at 90% of the maximum aerobic power, PMA). The following two experimental visits (#V4 and #V5) will replicate the tests described in #V3. However, during the constant load exercise, participants will breathe either ambient air or heliox (a mixture in which the nitrogen in the air is replaced by the inert gas helium) in a random order. During a final Experiential Visit (#V6), participants will replicate the "Medical Gas Administration" visit but the exercise will be interrupted when a similar amount of time/work as the ambient air condition is achieved.
Other: Air — Following the selection visit (#V0) to verify the inclusion and non-inclusion criteria, participants will make 2 visits (#V1 and #V2) including in particular a Respiratory Functional Exploration (EFR) and a triangular VO2 MAX estimation test in Ambient Air or Heliox conditions (depending on randomization).

SUMMARY:
It is generally accepted that the ventilatory system is not a limiting factor in physical exercise in terms of performance or exercise tolerance in healthy subjects. The ventilatory system would be oversized in relation to the stresses it has to cope with, even during maximum intensity exercise. However, some highly trained endurance athletes may be exceptions to this rule. A limitation of the expiratory flow is indeed sometimes found in these athletes, whose maximum values of ventilation can confront the mechanical limits of their ventilatory system. This phenomenon could be accentuated in elderly athletes (known as "master athletes") under the effect of structural and functional pulmonary alterations that accompany aging. Our hypothesis : What is the prevalence of exercise expiratory flow limitation in the master athlete and does it cause a decrease in physical performance via an acceleration of locomotor muscle fatigue?

ELIGIBILITY:
Inclusion Criteria:

* Non-smoker (active or passive) or ex-smoker of less than 5 pack-years and stopped for more than 10 years.
* No known significant chronic pathology.
* No symptoms suggesting a progressive pathology.
* No contraindication to physical exercise. Normal Pulmonary Functional Test (PFT).
* Participants affiliated to the social security system

Exclusion Criteria:

* Vulnerable persons as defined in Articles L. 1121-5 to L.1121-8 and L.1122-1-2 of the Public Health Code (e.g. persons deprived of liberty, minors, adults protected, etc.),
* Participants with a medical contraindication to sports practice,
* Cardiovascular, respiratory, neuromuscular and/or significant metabolic,
* Participants with declared pathology or medical treatment,
* Smoking or drug use,
* Significant chronic drug treatment,
* Lack of consent.
* Refusal to cooperate
* Recent rhino-bronchial infection (within last 4 weeks)
* Mental disability

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline severity of EFL during ergocycle endurance exercise | At inclusion and 3 months
  Force developed by the quadriceps muscle in response to percutaneous electrical stimulation of the femoral nerve

SECONDARY OUTCOMES:
Muscle activation level | At inclusion and 3 months
  estimated by measuring electromyographic (EMG) activity

CONTACTS AND LOCATIONS:
Overall Officials: Leroy Sylvie, Principal Investigator — Pneumologie, CHU de Nice
Locations (1):
- CHU de Nice, Nice, Alpes-maritimes, France

IPD SHARING:
Plan to Share IPD: No